CLINICAL TRIAL: NCT01047644
Title: Extended Interval Port Flushes: A Phase II Clinical Trial
Brief Title: Port Will be Flushed Every 3 Months Instead of Every 4-6 Wks, as Recommended by Port Manufacturer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Goetz Kloecker, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 09.0036
Record Dates: First submitted 2010-01-11; First posted 2010-01-13 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Complication of Catheter
Keywords: port; catheter; infusion; flush; cleanse; chemotherapy
MeSH Terms: conditions — Blushing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3-month flushing schedule (Experimental): 3-month port-flushing schedule
  Interventions: Other: Reduced port-flush schedule

INTERVENTIONS:
Other: Reduced port-flush schedule — 3-month port-flushing

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of port (PAC) flushes every 3 months rather than every four to six weeks.

It is routine practice to flush ports every four to six weeks, according to the manufacturer's recommendations, using salt solution followed heparin if needed. This study examines the effectiveness of port flushes at an alternative interval of 3 months, reducing the number of visits to the health-care provider.

DETAILED DESCRIPTION:
This is a phase II, non-blinded, non-inferiority prospective cohort trial of patients with ports (PAC) after a systemic therapy to evaluate the safety and effectiveness of PAC flushes in 3 months intervals. Patients with any type of cancer are eligible. The study will extend 1 year from enrollment of the last patient. Each enrolled patient will have his or her port flushed five times in 3 month intervals.

Patients will be enrolled after the completion of systemic therapy and after completion of the restaging follow up, which is the time period from 4 weeks to 3 months after discontinuation of the chemotherapy. Once patients are enrolled to extended interval PAC flushes, they will be followed for one year. At the end of the year patients will return to standard PAC flushes. If patients experience any PAC malfunction, it would be considered a PAC failure and the flushing will reverted back to the schedule recommended by the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

1. All patients 18 years and older with solid or hematological tumor who have a PAC after completion of curative intent treatment (Chemotherapy/Biotherapy)
2. Without active disease
3. Able to give informed consent

Exclusion Criteria:

1. Minors, prisoners
2. Previous PAC failure
3. Disease recurrence
4. Patients who had their PAC removed immediately following therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time to port complication | Every 3 months for 1 year
  The short-term endpoint is time to port complication (EFP- event free port-complication). The long term end point will be time to port failure requiring removal of the port (OAP - overal port failure) and will be used to determine the efficacy of port flushes every 3 months.

SECONDARY OUTCOMES:
Frequency and severity of toxicity | every three months
  Frequency and severity of toxicity will be monitored to describle incidence rates of toxicity.
Cost effectiveness | every three months
  Cost effectivenss will be estimated taking into consideration level of patient compliance and reduction in patient visits.

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, Principal Investigator — James Graham Brown Cancer Center, University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Diaz JA, Rai SN, Wu X, Chao JH, Dias AL, Kloecker GH. Phase II Trial on Extending the Maintenance Flushing Interval of Implanted Ports. J Oncol Pract. 2017 Jan;13(1):e22-e28. doi: 10.1200/JOP.2016.010843. Epub 2016 Oct 23. PMID 28084883
- See also: James Graham Brown Cancer Center, Louisville, KY — http://www.browncancercenter.org